CLINICAL TRIAL: NCT06205147
Title: Effects of Elastic Band Resistance Exercise on Muscle Strength and Depression in Hospitalized Elderly Patients.
Brief Title: Effects of Elastic Band Resistance Exercise on Muscle Strength and Depression in Hospitalized Elderly.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Piao-Yi Chiou, Associate Professor, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202306142RIND
Record Dates: First submitted 2023-10-24; First posted 2024-01-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Resistance Exercise; Muscle Weakness; Functional Decline
Keywords: resistance exercise; hospitalized elderly; muscle strength; depression; Functional decline
MeSH Terms: conditions — Muscle Weakness; Depression

STUDY DESIGN:
Intervention Model Description: Random control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short Falls Efficacy Scale International (Experimental): The Short Falls Efficacy Scale International (Short FES-I) consists of 7 questions. Scores range from a minimum of 7 points (no fear of falling) to a maximum of 28 points (severe fear of falling). Scores of 7 to 8 points indicate low concern about falling, 9 to 13 points indicate moderate concern about falling, and 14 to 28 points indicate high concern about falling.
  Interventions: Device: Elastic Band
- Geriatric Depression Scale, GDS 15 (Experimental): The assessment will be conducted within one week. Depressive symptoms in the elderly will be evaluated using a binary method, with answers of "yes" or "no." Questions 1, 5, 7, 11, and 13 should be answered with "no." Questions 2, 3, 4, 6, 8, 9, 10, 12, 14, and 15 should be answered with "yes." Each "yes" response is assigned 1 point, resulting in a total score of 15 points. Scores ranging from 0 to 6 indicate good emotional adjustment, scores from 7 to 10 indicate moderate emotional distress, and scores above 11 indicate severe emotional distress.
  Interventions: Device: Elastic Band

INTERVENTIONS:
Device: Elastic Band — Using the newly patented product, the Muscle Exercise and Falling Prevention Elastic Strap (Patent Certificate No. M585601), the procedure involves securing the elastic strap to a high-back chair to administer elastic band intervention exercises for patients.Guided by continuous contextual action demonstration videos, participants will engage in the elastic band resistance intervention twice a day, each session lasting 20 minutes, over a span of five days. These videos are designed to provide a continuous contextual demonstration, incorporating them within the video itself.

SUMMARY:
With improved a five-day intensive, low-resistance elastic band exercise program to evaluate its effectiveness in improving total muscle mass, upper and lower extremity muscle strength, self-perceived fear of falling, and depression among hospitalized elderly individuals. This study is a random control trial. Data collection includes elderly patient's total muscle mass, upper and lower extremity muscle strength, self-perceived fear of falling, and depression among hospitalized. The total muscle mass and upper and lower extremity muscle strength will be calculated in kilograms.

DETAILED DESCRIPTION:
Investigators have designed a five-day intensive, low-resistance elastic band exercise program to evaluate its effectiveness in improving total muscle mass, upper and lower extremity muscle strength, self-perceived fear of falling, and depression among hospitalized elderly individuals.

Investigators will enroll individuals aged 65 hospitalized elderly. participants will be randomly assigned to either the experimental or control group. The experimental group will undergo a five-day resistance exercise program using elastic bands, with two 20-minute sessions per day (totaling 200 minutes). The program aims to improve muscle mass and strength. Non-invasive instruments will be used to measure muscle mass and strength, and participants will complete self-report questionnaires on fear of fall and geriatric depression.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 65 years or older.
2. Anticipated hospital stay exceeding 7 days.
3. Able to follow instructions.
4. Four-limb muscle strength of at least three points, and grip strength measurements with a minimum of 26 kilograms for males and 18 kilograms for females.

Exclusion Criteria:

1. This includes individuals with cardiovascular diseases such as acute myocardial infarction, unstable angina, poorly controlled arrhythmias, complete atrioventricular block, acute heart failure, acute myocarditis, acute pericarditis, and other cardiac conditions.
2. Poorly controlled hypertension, with systolic blood pressure less than 90 mmHg or greater than 200 mmHg under medication.
3. Individuals hospitalized due to acute neurological injuries or conditions, such as epilepsy, stroke, or Parkinson's disease.
4. Diagnosed with cognitive impairment or Alzheimer's disease.
5. Those who require long-term ventilator support and are unable to participate in the program.
6. Individuals with impaired consciousness who cannot cooperate.
7. A Glasgow Coma Scale score of less than 12, or inability to correctly answer questions about person, time, place, or follow instructions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
total muscle mass and upper and lower extremity muscle strength | 20 minutes
  The changes in muscle mass and muscle strength will be measured before and after the intervention,The total muscle mass and upper and lower extremity muscle strength will be calculated in kilograms.

SECONDARY OUTCOMES:
Short Falls Efficacy Scale International Short FES | 20 minutes
  We will use the scale to measure changes in concerns about falling before and after the intervention.

OTHER OUTCOMES:
Geriatric Depression Scale, GDS 15. | 20 minutes
  The Geriatric Depression Scale (GDS-15) will be employed to measure changes in depressive symptoms among the elderly before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing of National Taiwan University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No